CLINICAL TRIAL: NCT00001272
Title: A Phase I Study of Taxol, Cisplatin, Cyclophosphamide and Granulocyte Colony-Stimulating Factor (G-CSF) in Previously Nontreated Ovarian Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 910232; 91-C-0232
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: Ovarian Neoplasms
Keywords: Adult; Cytotoxic Chemotherapy; Hematopoietic Growth Factor
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Paclitaxel

INTERVENTIONS:
Drug: taxol

SUMMARY:
This is a Phase I study which addresses the feasibility and toxicity of adding taxol to the two drug combination which now comprises the standard of care in newly diagnosed advanced stage ovarian cancer, cisplatin and cyclophosphamide. These drugs will be given in a dose intensive fashion with the colony-stimulating factor, G-CSF. Newly diagnosed patients with ovarian cancer will be treated with this regimen to determine the optimal dose of this combination. The pharmacokinetics of taxol and cisplatin DNA-adducts will be studied as well.

DETAILED DESCRIPTION:
This is a Phase I study which addresses the feasibility and toxicity of adding taxol to the two drug combination which now comprises the standard of care in newly diagnosed advanced stage ovarian cancer, cisplatin and cyclophosphamide. These drugs will be given in a dose intensive fashion with the colony-stimulating factor, G-CSF. Newly diagnosed patients with ovarian cancer will be treated with this regimen to determine the optimal dose of this combination. The pharmacokinetics of taxol and cisplatin DNA-adducts will be studied as well.

ELIGIBILITY:
All patients must have biopsy proven ovarian cancer as determined by evaluation in the Laboratory of Pathology, NCI.

Germ cell and borderline histologies are specifically excluded.

Patients must have FIGO stage III and IV disease, or FIGO Stage IIC disease with poorly differentiated histology, and will undergo attempted surgical debulking prior to the initiation of chemotherapy.

Prior chemotherapy or radiation therapy will make a patient ineligible.

Performance status: less than or equal to ECOG 2.

Patients must have the following end organ function:

No brain involvement.

No history of myocardial infarction, cardiac arrhythmias requiring

therapy, right bundle branch block with left anterior hemiblock, and left bundle branch block.

Renal function: creatinine clearance greater than or equal to 60 cc/min; patients with ureteral obstruction must have this corrected prior to starting therapy.

Hepatic function: normal coagulation parameters, serum transaminases within 3 times upper limit of normal.

Neurologic function: no preexisting dysfunction greater than grade 1 (exclusive of mild vibratory delay).

No recent history of active GI bleeding.

Hematologic parameters prior to starting cycle 1 of therapy: total granulocyte count greater than 2000 and platelet count greater than 100,000.

Patients may not have had prior history of invasive malignancy with the exception of nonmelanoma skin cancer curatively treated.

Patients must be able to give written informed consent and express a willingness to meet all of the expected requirements of the protocol.

Patients must be able to begin therapy within 8 weeks of staging laparotomy and should have a central venous catheter placed for infusion of chemotherapy.

All patients must be registered by calling the Orkand Corporation at 402-1732 between the hours of 8:30 AM and 5:00 PM; eligibility criteria will be queried.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1991-09; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States